CLINICAL TRIAL: NCT03248726
Title: Comparison of Single-dose (Morning) Low-volume Polyethylene Glycol Plus Bisacodyl Versus Split-dose Polyethylene Glycol for Bowel Preparation Efficacy in Patient Receiving Morning Colonoscopy
Brief Title: Comparing Single-dose Low-volume PEG Plus Bisacodyl vs. Split-dose PEG for Bowel Preparation in Morning Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: N201610042
Record Dates: First submitted 2017-05-31; First posted 2017-08-14 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Bowel Preparation
Keywords: Polyethylene Glycol; Bisacodyl; Colonoscopy; Bowel preparation; Ottawa bowel preparation scale
MeSH Terms: interventions — Polyethylene Glycols; Bisacodyl; klean prep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyethylene glycol and bisacodyl (Experimental): In order to decrease the dose and frequency of polyethylene glycol, we added bisacodyl at the night before examination to facilitate the action of polyethylene glycol given solely in the morning of examination.
  Interventions: Drug: Polyethylene glycol and bisacodyl
- Split-dose polyethylene glycol (Active Comparator): The standard regimen of polyethylene glycol was used in this group. The participant of this arm receives polyethylene glycol in the evening before examination and the morning of examination .
  Interventions: Drug: Split-dose polyethylene glycol

INTERVENTIONS:
Drug: Polyethylene glycol and bisacodyl — Intervention: Take 3 tablets (15mg) of stimulant laxatives Dulcolax® (bisacodyl) at 10pm the day before examination. Take two pack of osmotic laxative Klean-prep® powder (Polyethylene glycol) mixed with 2000ml water at 5am on the morning of examination.
  Other Names: Dulcolax®; Klean-prep®
  Arms: Polyethylene glycol and bisacodyl
Drug: Split-dose polyethylene glycol — Take two pack of Klean-prep® powder mixed with 2000ml water at 6pm before the day of examination, and take another two pack of osmotic laxative Klean-prep® powder mixed with 2000ml water at 5am on the examination day.
  Other Names: Klean-prep®
  Arms: Split-dose polyethylene glycol

SUMMARY:
Colonoscopy is the best method to detect colorectal cancer and colonic polyps. Studies showed that adenoma detection rate positive correlation with good bowel preparation which makes bowel preparation an important issue. Hence, investigators conduct a clinical trial about adding another laxative agent to morning single dose low-volume PEG. To see if this new regimen could have non-inferior efficacy and lower life/sleep impact compared with standard regimen.

DETAILED DESCRIPTION:
Colorectal cancer incidence rate has increased in recently years, and colorectal cancer has come to the top of cancer incidence ranking of Taiwan. Colonoscopy is the best method to detect colorectal cancer and colonic polyps. Studies showed that adenoma detection rate positive correlation with good bowel preparation. That makes bowel preparation an important issue. Polyethylene Glycol (PEG) is widely used for bowel preparation for it efficacy and safety. However, there are many different adjunctive, dose, timing of administration in PEG preparation. Some may decrease patient tolerability due to large fluid volume, and some may influence patient's life and sleep quality when performing bowel preparation. Here, investigators conduct a clinical trial about adding another laxative agent to morning single dose low-volume PEG. To see if this new regimen could have non-inferior efficacy and lower life/sleep impact compared with standard regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-70 years.
* Out-patient department ambulatory patient.
* Patients who have indications to receive colonoscopy.

Exclusion Criteria:

* Age is under 20 or over 70
* Have severe renal impairment (hemodialysis or eGFR<30).
* Have severe congestive heart failure (NYHAⅢorⅣ).
* Pregnant or lactating, or women is under oral contraceptive.
* Have history of bowel obstruction or resection, known or suspected gastroparesis acute gastric/intestinal ulcer, toxic colitis or megacolon
* Be allergic to polyethylene glycol (PEG) or bisacodyl.
* Have severe constipation ( ≤ 1 bowel movement per week).
* Patient who has Phenylketonuria.
* Refuse to sign consent to the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The Ottawa Bowel Preparation Scale | Within 24 hours after colonoscopy
  Examiner will fill a case report form out after performing a colonoscopy. Score below or equal to 6 will be classified as "good preparation".

SECONDARY OUTCOMES:
Life disturbance | 30 minutes before patient receive colonoscopy
  Evaluate patients life disturbance with a questionnaire before performing a colonoscopy. The questionnaire including side effect, sleep quality, interference of life/work, and tendency of same bowel preparation method at next colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Cheng Huang, Bachelor, Principal Investigator — Gastroenterology division, Internal Medicine Department, Wanfang Hospital
Locations (1):
- Wanfang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No